CLINICAL TRIAL: NCT04584359
Title: Comparasion of the Effects of Osteopathic Manipulations and Muscle Training on the Myoelectric Activity of the Pelvic Floor in Women With Stress Urinary Incontinence: a Randomized Controlled Trial.
Brief Title: Effects of Osteopathic Manipulations and Muscle Training on the Myoelectric Activity of the Pelvic Floor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giselle Notini Arcanjo (Other)
Responsible Party: Sponsor-Investigator, Giselle Notini Arcanjo, Principal Investigator, University of Trás-os-Montes and Alto Douro
Organization: University of Trás-os-Montes and Alto Douro (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Utras1
Record Dates: First submitted 2020-08-24; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Urinary Incontinence
Keywords: pelvic floor training; osteopathy; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Heimlich Maneuver

STUDY DESIGN:
Intervention Model Description: This study randomized 40 women with symptoms of stress uriray incontinence who were divided into four intervention groups of ten women each (G1: only the high velocity, low amplitude manipulation for the sacroiliac joint and T10-L2; G2: global osteopathic protocol with myofascial, visceral, and articular techniques; G3: pelvic floor muscle training; and G4: control).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HVLA techiniques (G1) (Experimental): Performed with thrust (also known as HVLA) in the sacroiliac joint and T10-L2 level
  Interventions: Other: HVLA; Other: global osteopathic protocol
- Global osteopathic protocol (G2) (Experimental): Several elements were emphasized - myofascial, bone, and visceral.
  Interventions: Other: global osteopathic protocol
- Pelvic floor muscle training (G3) (Experimental): Muscle Training for four weeks, with a weekly face-to-face visit lasting 10-20 minutes.
  Interventions: Other: pelvic floor muscle training
- Control group (G4) (No Intervention): No intervention and was simply evaluated and re-evaluated.

INTERVENTIONS:
Other: HVLA — High velocity, low amplitude manipulation for the sacroiliac joint and T10-L2. The interventions were performed once a week for four weeks by a physiotherapist with a degree in in osteopathy and ten years of clinical experience. Each visit lasted about 5 minutes.
  Other Names: thrust
  Arms: HVLA techiniques (G1)
Other: global osteopathic protocol — Myofascial, visceral, and articular techniques. Complete treatment in order to restore and rebalance internal tensions and improve the visceral mobility: muscle inhibition techniques for the psoas muscle; deep massage in the obturator foramen; stretching for the greater omentum; lift of the uterus, ovary, and bladder ; abdominal maneuver; and thrust of sacroiliac joint and T12-L1. The interventions were performed once a week for four weeks by a physiotherapist with a degree in in osteopathy and ten years of clinical experience. Each visit lasted about 15 minutes.
  Arms: Global osteopathic protocol (G2); HVLA techiniques (G1)
Other: pelvic floor muscle training — Pelvic floor muscle training for four weeks, with a weekly face-to-face visit lasting 10-20 minutes. In this intervention, participants were instructed to perform three sequences of exercises: contractions and relaxations (three seconds of sustained contractions and six seconds of rest), ten sustained contractions (ten seconds of sustained contractions and 20 seconds of rest), and five contractions associated with a cough. These exercises were performed in the standing, sitting, and lying positions
  Arms: Pelvic floor muscle training (G3)

SUMMARY:
The objective of this study was to compare the effects of four different interventions on pelvic floor muscle electromyographic activity in women with stress urinary incontinece: i) a global osteopathic protocol (myofascial, visceral, and articular techniques), ii) one manipulation technique (high velocity, low amplitude (HVLA)/thrust) of the sacroiliac joint and T10-L2, iii) Pelvic Floor Muscle training, and iv) a control group with no intervention. The hypothesis is that the global osteopathic protocol and HVLA technique can increase pelvic floor muscle electromyographic activity to a level greater than or equal to the standard care established in the literature (pelvic floor muscle training).

DETAILED DESCRIPTION:
Participants represented a convenience sample and were recruited from hospitals, urogynecology doctors' clinics, invitations via social networks, gyms, clubs, and sports consultants. Women had to be between 30 and 60 years old and report symptoms of urine loss due to exertion in the last six months.The participants were randomly allocated into four groups (G1 = intervention using an HVLA/thrust technique for the sacroiliac and T10-L2 joints, G2 = global osteopathic protocol, G3 = PFT, and G4 = control) by a blinded researcher with a spreadsheet of random numbers.The primary outcome measure was surface electromyography (EMG) performed at five different times: before the intervention and immediately, 30 minutes, 60 minutes, and four weeks after. This evaluation was performed by a physiotherapist with ten years of experience in urogynecology and expertise in PFM electromyographic evaluation who was blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of urine loss due to exertion in the last six months.

Exclusion Criteria:

* urgent or mixed urinary incontinency
* overactive bladder
* neurological disorder
* urinary or anal infection
* urogenital atrophy
* pelvic organ prolapse grade 3 or 4
* sensory pathways and motor not intact
* spine fracture

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
electromyographic activity | Change from baseline versus immediately post-intervention
  The primary outcome measure will be the RMS (root means square) collected by surface. First, the basal tonus activity of PFM was recorded for 20 seconds; participants were instructed to avoid any body movements or speech. Next, the participants performed two fast and consecutive contractions (three seconds each) and relaxed for ten seconds (test for phasic fibers). Third, participants were told to sustain the contraction for ten seconds, followed by a ten-second rest (test for tonic fibers). Finally, the myoelectrical activity was captured during a cough to assess PFM reflex contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle N Arcanjo, Principal Investigator — Tras dos Montes Alto Douro University
Locations (1):
- Giselle Notini Arcanjo, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams, P., Cardozo, L., Wagg, A., Wein, A. (Eds). (2017). Incontinence. 6th Edition. ICI-ICS. International Continence Society, Bristol UK.
- [Background] Fernandes, W.V.B., Bicalho, E.S., Capote, A.E., Manffra E.F. (2016). Duration of the effects of spinal manipulation on pain intensity and electromyographic activity of paravertebral parts of individuals with chronic mechanical low back pain. Fisioterapia Pesquisa, 23(2),155-62
- [Background] Felicíssimo, M.F., Carneiro, M.M., Souza, E.L.B.L. de, Alipio, V.G., Franco, M.R.C., Silva, R. G. O., Filho, A.L.S. (2016). Fatores limitadores à reabilitação da musculatura do assoalho pélvico em pacientes com incontinência urinária de esforço. Acta Fisiátrica, 14(4), 233-236
- [Background] Franke H, Hoesele K. Osteopathic manipulative treatment (OMT) for lower urinary tract symptoms (LUTS) in women. J Bodyw Mov Ther. 2013 Jan;17(1):11-8. doi: 10.1016/j.jbmt.2012.05.001. Epub 2012 Jun 17. PMID 23294678
- [Background] Glazer, H. I.; Hacad, C. R. (2012). The Glazer Protocol: Evidence-Based Medicine Pelvic Floor Muscle (PFM) Surface Electromyography (SEMG). Biofeedback, 40(2), 75-79
- [Background] Herzog W. The biomechanics of spinal manipulation. J Bodyw Mov Ther. 2010 Jul;14(3):280-6. doi: 10.1016/j.jbmt.2010.03.004. PMID 20538226
- [Background] Lopez, D. Osteopathy for Urologic and Pelvic Health. In: Chughtai, B.; Stein, A. Espinosa, G. (2017). Healing In Urology Clinical Guidebook to Herbal and alternative therapies, cap 10, pp. 209-221
- [Background] Palma, P. C. R. (2009). Aplicações clínicas das técnicas fisioterapêuticas nas disfunções miccionais e do assoalho pélvico. Campinas, SP, Personal Link Comunicações
- [Background] Resende, A. P. M., Nakamura, M. U., Ferreira, E. A. G., Petricelli, C. D., Alexandre, S. M., Zanetti, M. R. D. (2011). Evaluation of female pelvic floor muscles using surface electromyography: literature review. Fisioterapia e Pesquisa, 18(3), 292-297
- [Result] de Andrade RL, Bo K, Antonio FI, Driusso P, Mateus-Vasconcelos ECL, Ramos S, Julio MP, Ferreira CHJ. An education program about pelvic floor muscles improved women's knowledge but not pelvic floor muscle function, urinary incontinence or sexual function: a randomised trial. J Physiother. 2018 Apr;64(2):91-96. doi: 10.1016/j.jphys.2018.02.010. Epub 2018 Mar 21. PMID 29574170
- [Result] de Almeida BS, Sabatino JH, Giraldo PC. Effects of high-velocity, low-amplitude spinal manipulation on strength and the basal tonus of female pelvic floor muscles. J Manipulative Physiol Ther. 2010 Feb;33(2):109-16. doi: 10.1016/j.jmpt.2009.12.007. PMID 20170776
- [Result] Alves JO, Luz STD, Brandao S, Da Luz CM, Jorge RN, Da Roza T. Urinary Incontinence in Physically Active Young Women: Prevalence and Related Factors. Int J Sports Med. 2017 Nov;38(12):937-941. doi: 10.1055/s-0043-115736. Epub 2017 Sep 26. PMID 28950397
- [Result] Araujo MP, Sartori MGF, Girao MJBC. Athletic Incontinence: Proposal of a New Term for a New Woman. Rev Bras Ginecol Obstet. 2017 Sep;39(9):441-442. doi: 10.1055/s-0037-1605370. Epub 2017 Jul 20. No abstract available. PMID 28728191
- [Result] Batista RL, Franco MM, Naldoni LM, Duarte G, Oliveira AS, Ferreira CH. Biofeedback and the electromyographic activity of pelvic floor muscles in pregnant women. Rev Bras Fisioter. 2011 Sep-Oct;15(5):386-92. doi: 10.1590/s1413-35552011005000026. Epub 2011 Oct 14. English, Portuguese. PMID 22002190
- [Result] Bertotto A, Schvartzman R, Uchoa S, Wender MCO. Effect of electromyographic biofeedback as an add-on to pelvic floor muscle exercises on neuromuscular outcomes and quality of life in postmenopausal women with stress urinary incontinence: A randomized controlled trial. Neurourol Urodyn. 2017 Nov;36(8):2142-2147. doi: 10.1002/nau.23258. Epub 2017 May 16. PMID 28508398
- [Result] Cuthbert SC, Rosner AL. Conservative chiropractic management of urinary incontinence using applied kinesiology: a retrospective case-series report. J Chiropr Med. 2012 Mar;11(1):49-57. doi: 10.1016/j.jcm.2011.10.002. PMID 22942842
- [Result] Dasikan Z, Ozturk R, Ozturk A. Pelvic floor dysfunction symptoms and risk factors at the first year of postpartum women: a cross-sectional study. Contemp Nurse. 2020 Apr;56(2):132-145. doi: 10.1080/10376178.2020.1749099. Epub 2020 Apr 7. PMID 32216721
- [Result] Haavik H, Murphy BA, Kruger J. Effect of Spinal Manipulation on Pelvic Floor Functional Changes in Pregnant and Nonpregnant Women: A Preliminary Study. J Manipulative Physiol Ther. 2016 Jun;39(5):339-347. doi: 10.1016/j.jmpt.2016.04.004. Epub 2016 May 6. PMID 27157677
- [Result] Horton, R.C. (2015). The anatomy, biological plausibility and efficacy of visceral mobilization in the treatment of pelvic ﬂoor dysfunction. Journal of Pelvic, Obstetric and Gynaecological Physiotherapy, 117, 5-18
- [Result] Lopes MH, Costa JN, Lima JL, Oliveira LD, Caetano AS. Pelvic floor rehabilitation program: report of 10 years of experience. Rev Bras Enferm. 2017 Jan-Feb;70(1):231-235. doi: 10.1590/0034-7167-2016-0257. English, Portuguese. PMID 28226063
- [Result] Ponzoni, L. de C.; Valentin E.K.; Carrerette F.B.; Damião, R. (2019). Musculoskeletal osteopathic manipulative treatment in women with uncomplicated urinary incontinence. Fisioterapia Brasil, 20(2), 230-8
- [Result] Santos MD, Palmezoni VP, Torelli L, Baldon VSP, Sartori MGF, Resende APM. Evaluation of pelvic floor muscle strength and its correlation with sexual function in primigravid and non-pregnant women: A cross-sectional study. Neurourol Urodyn. 2018 Feb;37(2):807-814. doi: 10.1002/nau.23353. Epub 2017 Aug 1. PMID 28762553
- [Result] Tettambel MA. An osteopathic approach to treating women with chronic pelvic pain. J Am Osteopath Assoc. 2005 Sep;105(9 Suppl 4):S20-2. PMID 16249362
- [Result] Thomaz RP, Colla C, Darski C, Paiva LL. Influence of pelvic floor muscle fatigue on stress urinary incontinence: a systematic review. Int Urogynecol J. 2018 Feb;29(2):197-204. doi: 10.1007/s00192-017-3538-6. Epub 2017 Dec 20. PMID 29264615
- [Result] Celiker Tosun O, Kaya Mutlu E, Ergenoglu AM, Yeniel AO, Tosun G, Malkoc M, Askar N, Itil IM. Does pelvic floor muscle training abolish symptoms of urinary incontinence? A randomized controlled trial. Clin Rehabil. 2015 Jun;29(6):525-37. doi: 10.1177/0269215514546768. Epub 2014 Aug 20. PMID 25142280